CLINICAL TRIAL: NCT03235154
Title: Bridging Care to HCV Treatment Among Opiate Dependent Patients on Buprenorphine/Naloxone Maintenance Therapy: A Pilot Study of Treating HCV With Epclusa at a Psychiatrist-staffed Outpatient Addiction Clinic
Brief Title: A Pilot Study of Treating HCV at a Psychiatrist-staffed Outpatient Addiction Clinic
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Community Research Initiative of New England (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-05
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C, Chronic; Hepatitis C; Opiate Dependence
Keywords: HCV; Suboxone; Epclusa; psychiatrist
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C; Opioid-Related Disorders | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Other): In this open label, single arm study, all subjects will receive the intervention as prescribed by psychiatrists in the office based opiate addition treatment program.
  Interventions: Drug: sofosbuvir/velpatasvir

INTERVENTIONS:
Drug: sofosbuvir/velpatasvir — 12 week treatment with once daily sofosbuvir/velpatasvir fixed dose combination therapy. Tablets are formulated with 400mg sofosbuvir and 100mg velpatasvir in pink, diamond-shaped, film coated tablets.

SUMMARY:
The main purpose of this pilot study is to investigate the safety, effectiveness and tolerability of the study medication in the treatment of people with chronic hepatitis C virus infection who regularly attend a psychiatrist-staffed clinic for opiate addiction treatment.

DETAILED DESCRIPTION:
An estimated 3.2 million people in the United States are currently infected with hepatitis C virus (HCV). Since 1990, when the US introduced screening of the blood supply for HCV, injection drug use has been the primary mode of HCV transmission in the United States. It is widely recognized that addressing the HCV epidemic among people who inject drugs (PWID) depends on increasing access to: 1) clean injection equipment; 2) opiate substitution therapy (OST); 3) curative HCV treatment; and 4) assistance with comorbid psychiatric conditions and social issues (Robaeys, C et al, 2013).

Nevertheless, access to HCV treatment among current and former injection drug users is thought to be limited by several factors including: 1) insufficient number of infectious disease and gastroenterology providers and 2) provider and third-party payor concerns about adherence to medication and the risk of reinfection (Aspinall, EJ et al, 2013). Strategies to increase access among current and former injection drug users to direct acting antiviral drugs are urgently needed. The purpose of the current study is to assess the impact of co-treating chronic hepatitis C infection and opiate dependence within the context of an outpatient addiction clinic staffed by psychiatrists. The beneficial impact of co-treating opiate dependence and an infectious illness has been demonstrated in the case of HIV infection. Altice and colleagues conducted an observational study of HIV-infected opiate-dependent patients who were offered OST with buprenorphine/naloxone at 10 different HIV clinics. Subjects initiating buprenorphine/naloxone were more likely to initiate or remain on ART (antiretroviral therapy) (Altice, 2011).

The Extension for Community Healthcare Outcomes (ECHO) program has demonstrated that with proper training and mentorship, primary care providers with no prior experience in managing HCV are able to treat the disease effectively (Arora et al, 2011). Since the publication of the ECHO study, the treatment of HCV has become considerably less complicated due to the widespread availability of safe, highly effective single tablet regimens, such as Epclusa. The investigators believe that treatment of HCV is now well within the grasp of physicians and other healthcare providers without training in internal or family medicine.

This single arm pilot study will assess HCV treatment with Epclusa at an outpatient addiction clinic staffed by psychiatrists. The investigators hypothesize that with proper training and mentorship, psychiatrists who are also a licensed buprenorphine/naloxone providers will be able to effectively assess liver health and treat chronic hepatitis C infection with Epclusa. Further, the investigators hypothesize that patients with chronic hepatitis C infection on buprenorphine/naloxone maintenance therapy who are treated for HCV by a psychiatrist during regularly scheduled visits to an addiction clinic will have high rates of adherence to HCV treatment and achieve SVR12 (sustained virologic response, 12 weeks post-treatment).

Given that subjects will receive standard of care evaluation and treatment for their chronic hepatitis C infection, the investigators believe that study participation poses minimal risk. Indeed, The investigators believe that subjects will benefit from improved access to this important treatment which will be provided at a convenient location by a known physician under the guidance of an infectious disease physician with extensive experience treating HCV infection.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age ≥ 18 years
3. Confirmation of chronic HCV infection as documented by a positive HCV antibody test at least 6 months prior to the Baseline/Day 1 visit and positive HCV RNA test at screening
4. HCV genotype 1, 2, 3, 4, 5 or 6
5. In stable remission from opiate use on buprenorphine/naloxone for at least 12 weeks
6. Within the following laboratory parameters as assessed at the screening visit:

   1. HCV RNA quantifiable
   2. Screening rhythm strip without bradycardia (heart rate > 60 or, if on beta blocker, > 55 BPM)
   3. Alanine Aminotransferase (ALT) ≤ 10 x ULN (upper limit of normal)
   4. Aspartate Aminotransferase (AST) ≤ 10 x ULN
   5. Direct bilirubin ≤ 1.5 x ULN
   6. Platelets > 60,000
   7. Hemoglobin A1C (HbA1c) ≤ 10%
   8. Creatinine clearance ≥ 30 mL/min, as calculated by the Cockcroft-Gault equation
   9. Albumin ≥ 3g/dL
   10. International Normalized Ratio (INR) ≤ 1.5 x ULN or on an anticoagulant regimen affecting INR
7. Female subject is eligible to enter if it is confirmed that she is:

   1. Not pregnant or nursing
   2. Not of childbearing potential (i.e. s/p hysterectomy, oophorectomy or has medically documented ovarian failure, or are postmenopausal women > 50 years of age with cessation of menses for 12 months or greater) OR Of childbearing potential with a negative serum pregnancy test within 2 weeks of screening, a negative urine pregnancy test on Day 1, and a commitment to either abstain from intercourse or consistently use an acceptable method of birth control (Appendix 4) in addition to condom use by her male partner(s) from the date of screening until 30 days after the last dose of study drug
8. All male study participants must agree to consistently and correctly use condoms with their female partner(s) and their female partner(s) must agree to use an acceptable method of birth control (listed) from the date of screening until 90 days after the last dose of study drug
9. Male subjects must refrain from sperm donation from the date of screening until 90 days after the last dose of study drug
10. Subject must be in generally good health, with the exception of HCV, in the opinion of the Sponsor-Investigator or Sub-Investigator(s)
11. Subject must be able to comply with dosing instructions for study drug administration and able to complete the study visits, including all required post-treatment visits

Exclusion Criteria:

1. Presence of decompensated cirrhosis as defined by encephalopathy, ascites, or a history of a variceal bleed
2. Prior treatment with direct acting antiviral hepatitis C medications
3. Positive urine drug toxicity test at screening (except for cannabinoids and prescribed medications)
4. Absence of buprenorphine in urine sample at screening
5. Currently pregnant or breastfeeding female
6. Detectable HIV RNA > 50 copies/ml (co-infected subjects with suppressed viral load are eligible for participation)
7. Use of any prohibited concomitant medication within 28 days prior to day 1
8. Chronic use of systemically administered immunosuppressive agents
9. Difficulty with blood collection or poor venous access
10. History of solid organ transplantation
11. Known significant allergy to sofosbuvir or velpatasvir
12. Current chronic liver disease of a non-HCV etiology (including hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency)
13. Active Hepatitis B virus (HBV) infection defined as either a positive HBV surface antigen test or a positive test for HBV DNA. (Subjects who are positive for HBV core antibody but negative for Hepatitis B surface antibody, surface antigen, and DNA ARE eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy E Colson, MD MPH, Principal Investigator — Community Research Initiative of New England
Locations (1):
- Cambridge Health Alliance Outpatient Addiction Services, Somerville, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altice FL, Bruce RD, Lucas GM, Lum PJ, Korthuis PT, Flanigan TP, Cunningham CO, Sullivan LE, Vergara-Rodriguez P, Fiellin DA, Cajina A, Botsko M, Nandi V, Gourevitch MN, Finkelstein R; BHIVES Collaborative. HIV treatment outcomes among HIV-infected, opioid-dependent patients receiving buprenorphine/naloxone treatment within HIV clinical care settings: results from a multisite study. J Acquir Immune Defic Syndr. 2011 Mar 1;56 Suppl 1(Suppl 1):S22-32. doi: 10.1097/QAI.0b013e318209751e. PMID 21317590
- [Background] Arora S, Thornton K, Murata G, Deming P, Kalishman S, Dion D, Parish B, Burke T, Pak W, Dunkelberg J, Kistin M, Brown J, Jenkusky S, Komaromy M, Qualls C. Outcomes of treatment for hepatitis C virus infection by primary care providers. N Engl J Med. 2011 Jun 9;364(23):2199-207. doi: 10.1056/NEJMoa1009370. Epub 2011 Jun 1. PMID 21631316
- [Background] Robaeys G, Grebely J, Mauss S, Bruggmann P, Moussalli J, De Gottardi A, Swan T, Arain A, Kautz A, Stover H, Wedemeyer H, Schaefer M, Taylor L, Backmund M, Dalgard O, Prins M, Dore GJ; International Network on Hepatitis in Substance Users. Recommendations for the management of hepatitis C virus infection among people who inject drugs. Clin Infect Dis. 2013 Aug;57 Suppl 2:S129-37. doi: 10.1093/cid/cit302. PMID 23884061
- [Background] Aspinall EJ, Corson S, Doyle JS, Grebely J, Hutchinson SJ, Dore GJ, Goldberg DJ, Hellard ME. Treatment of hepatitis C virus infection among people who are actively injecting drugs: a systematic review and meta-analysis. Clin Infect Dis. 2013 Aug;57 Suppl 2:S80-9. doi: 10.1093/cid/cit306. PMID 23884071

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm
Started | 11
Completed Epclusa. Treatment | 8
12-wk Post-treatment HCV RNA Measured | 7
Completed | 7
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Intervention: 12-week Epclusa Treatment
Arm/Group | Single Arm Intervention
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 48 [25 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11
Co-morbid axis 1 diagnosis present [Count of Participants; unit: Participants] — The presence of a co-morbid axis 1 diagnosis was confirmed by the treating psychiatrist. Axis 1 diagnoses refer to major mental disorders including mood disorders, anxiety disorders and schizophrenia/psychotic disorders
  Participants | 11
HCV (hepatitis C virus) RNA [Mean (Full Range); unit: IU/ml] | 2,662,207 [29384 to 10408895]
Baseline FibroSure fibrosis stage [Count of Participants; unit: Participants] — The level of liver fibrosis was determined by the FibroSure HCV blood test which uses a combination of six serum markers plus age and gender in a patented algorithm to generate a measure of fibrosis. The stages of fibrosis range from 0 (no fibrosis) to 4 (liver cirrhosis). Stage F1 refers to portal fibrosis, stage F2 to bridging fibrosis with few septa, and stage F3 to bridging fibrosis with many septa.
  Participants
    F0 | 6
    F1 | 2
    F2 | 0
    F3 | 1
    F4 | 0
    Unknown | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response at 12 Weeks Post Treatment (SVR-12)
Description: To assess the effectiveness of HCV treatment with velpatasvir/sofosbuvir administered by psychiatrist/licensed buprenorphine/naloxone providers during regularly scheduled visits to an outpatient addiction clinic for buprenorphine/naloxone replacement therapy and mental healthcare, as measured by percentage of patients achieving SVR-12 (defined as HCV RNA < lower limit of quantification (LLOQ) 12 weeks after discontinuation of study treatment),
Time Frame: This outcome measure will be assessed for each participant 12 weeks after completion of a 12 week course of treatment
Population: subjects who completed Epclusa treatment and had HCV RNA measured 12 weeks after completion of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Health-Related Quality of Life
Description: Change in mean score on 5-point LIkert Scale to statement "My Health is Excellent" (1=definitely true, 5=definitely false) from baseline and 12 weeks post-treatment
Time Frame: Baseline and 12 weeks post treatment
Population: Subjects who completed questionnaire at baseline and 12 weeks after completion of treatment
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Single Arm Intervention: Subjects who completed baseline and 12-week post treatment questionnaire
Arm/Group | Single Arm Intervention
Number analyzed (Participants) | 7
score on a scale | -0.44 [-1 to 0]

3. Secondary Outcome: Adherence to Study Treatment
Description: To assess adherence to velpatasvir/sofosbuvir therapy among participants administered treatment in the context of visits to an outpatient addiction clinic for buprenorphine/naloxone replacement therapy and mental health care.
Time Frame: This outcome measure will be assessed for each participant during a 12 week course of study treatment.
Population: The 8 subjects who completed treatment
Measure: Mean (Full Range); unit: % of prescribed doses taken
Arm/Group | Single Arm Intervention
Number analyzed (Participants) | 8
% of prescribed doses taken | 94 [83.7 to 100]
Statistical Analysis 1: Comparison: Single Arm Intervention; This was a single arm intervention study with a very small number of participants. Therefore, only descriptive statistics are provided; Test type: Other — There was no comparator arm in this small single arm study; No confidence intervals around point estimates provided given very small number of participants; No confidence intervals around point estimates provided given very small number of participants

ADVERSE EVENTS:
Time Frame: From study entrance through treatment period
Arm/Group | Single Arm Intervention
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Intervention (N=11)
Altered Mental Status (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Visual Hallucination (Nervous system disorders) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Intervention (N=11)
GI distress (Gastrointestinal disorders) | 2
Fatigue (Nervous system disorders) | 1
Scabies (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT03235154/Prot_SAP_001.pdf
  • Informed Consent Form: ICF for patients (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/54/NCT03235154/ICF_002.pdf
  • Informed Consent Form: ICF for providers (2017-05-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03235154/ICF_003.pdf